CLINICAL TRIAL: NCT02516527
Title: A Phase 1 Dose Escalation Study of the Safety, Tolerability, and Pharmacokinetics of Ipilimumab in Chinese Subjects With Select Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: CA184-247
Record Dates: First submitted 2015-07-03; First posted 2015-08-06 (Estimated); Last update posted 2020-05-01 (Actual); Status verified 2020-04

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma | interventions — Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Induction Phase:Ipilimumab (Experimental): Ipilimumab dose as specified
  Interventions: Drug: Ipilimumab
- Maintenance Phase:Ipilimumab (Experimental): Ipilimumab dose as specified
  Interventions: Drug: Ipilimumab

INTERVENTIONS:
Drug: Ipilimumab

SUMMARY:
The purpose of this study is to determine whether ipilimumab is effective in the treatment of select advanced (unresectable, metastatic, or recurrent) solid tumors in Chinese subjects.

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com.

Inclusion Criteria:

* Subjects with the following advanced solid tumors; metastatic or recurrent
* Must have measurable/non-measurable lesion per Response Evaluation Criteria in Solid Tumors (RECIST v1.1) criteria.
* Subjects have ability to comply with treatment, procedures and pharmacokinetics (PK) sample collection and the required study follow-up
* Chinese women and men, ages 18 years or older

Exclusion Criteria:

* Subjects with brain metastases are excluded unless clinically stable for more than 4 weeks at the time of randomization as determined by the investigator
* Subjects with ocular melanoma are excluded
* Any other malignancy from which the subject has been free of disease for less than two years, with the exception of adequately treated and cured basal or squamous cell skin cancer, superficial bladder cancer, or carcinoma in situ of the cervix
* History of, or currently active, autoimmune diseases, including but not limited to inflammatory bowel disease, rheumatoid arthritis, autoimmune hepatitis, systemic sclerosis (scleroderma and variants), systemic lupus erythematosus, autoimmune vasculitis, autoimmune neuropathies (eg, Guillain-Barre syndrome). Vitiligo is not excluded
* Any current or history of immunodeficiency, splenectomy, or splenic radiation

Other protocol defined inclusion/exclusion criteria could apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2015-10-16 (Actual); Primary Completion 2018-09-20 (Actual); Study Completion 2018-09-20 (Actual)

PRIMARY OUTCOMES:
The safety of ipilimumab measured by the occurrence of adverse events, serious adverse events, adverse events leading to discontinuation and deaths | Up to 90 days post discontinuation of dosing
The tolerability of ipilimumab measured by the occurrence of adverse events, serious adverse events, adverse events leading to discontinuation and deaths | Up to 90 days post discontinuation of dosing
Identify dose limiting toxicities in Chinese subjects with select advanced (unresectable, metastatic, or recurrent) solid tumors measured by the occurrence of adverse events, serious adverse events, adverse events leading to discontinuation, and deaths | Up to 90 days post discontinuation of dosing

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Ma Y, Fang W, Zhao H, Bathena SP, Tendolkar A, Sheng J, Zhang L. A Phase I Dose Escalation Study of the Safety, Tolerability, and Pharmacokinetics of Ipilimumab in Chinese Patients with Select Advanced Solid Tumors. Oncologist. 2021 Apr;26(4):e549-e566. doi: 10.1002/onco.13577. Epub 2020 Nov 11. PMID 33105036
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/investigator-inquiry-form.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm